CLINICAL TRIAL: NCT01249482
Title: Symptom Assessment for Patients With Gastro-esophageal Reflux Disease Receiving Helicobacter Pylori Eradication
Brief Title: Symptom Assessment for GERD Patients Receiving H. Pylori Eradication
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yi-Chia Lee, National Taiwan University Hospital
Other Study IDs: 201008001M
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-11

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Helicobacter pylori; reflux; acid rebound
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Late eradication: Group B (n=100) will be given rabeprazole 20 mg qd for 8 weeks and discontinued for 2 weeks. Then, H. pylori eradication with triple therapy will be given for one week, followed by rabeprazole 20 mg qd for 7 weeks.
- Negative HP: For patients with negative H. pylori infection (n=100), proton-pump inhibitor with rabeprazole 20 mg qd will be given for 8 weeks and discontinued.
- Early eradication: Group A (n=100) will be given initial H. pylori eradication with triple therapy for one week, followed by proton-pump inhibitor with rabeprazole 20 mg qd for 7 weeks.

SUMMARY:
Background: Rebound acid hypersecretion and acid-related symptoms after discontinuation of proton-pump inhibitor has been reported in previous studies. In patients with concurrent gastro-esophageal reflux disease and Helicobacter pylori infection, whether eradication of Helicobacter pylori (H. pylori)will aggravate acid-related symptoms after discontinuation of proton-pump inhibitor remains elusive Objective: This study aims to investigate the incidence and severity of acid-related symptoms after discontinuation of proton-pump inhibitor in reflux patients receiving H. pylori eradication.

DETAILED DESCRIPTION:
Background: Rebound acid hypersecretion and acid-related symptoms after discontinuation of proton-pump inhibitor has been reported in previous studies. In patients with concurrent gastro-esophageal reflux disease and Helicobacter pylori infection, whether eradication of H. pylori will aggravate acid-related symptoms after discontinuation of proton-pump inhibitor remains elusive Objective: This study aims to investigate the incidence and severity of acid-related symptoms after discontinuation of proton-pump inhibitor in reflux patients receiving H. pylori eradication Patients and methods: Consecutive reflux patients documented by validated questionnaires (GerdQ) and upper endoscopy will be enrolled from the outpatient clinic. After determination of H. pylori status by urea breath test, those with positive H. pylori infection will be randomized into two groups. Group A (n=100) will be given initial H. pylori eradication with triple therapy for one week, followed by proton-pump inhibitor (PPI) with rabeprazole 20 mg qd for 7 weeks. Group B (n=100) will be given rabeprazole 20 mg qd for 8 weeks and discontinued for 2 weeks. Then, H. pylori eradication with triple therapy will be given for one week, followed by rabeprazole 20 mg qd for 7 weeks. For patients with negative H. pylori infection (n=100), proton-pump inhibitor with rabeprazole 20 mg qd will be given for 8 weeks and discontinued. The incidence and severity of acid-related symptoms will be evaluated with GerdQ at 2 weeks after discontinuation of PPI. The impact of H. pylori infection and H. pylori eradication on the incidence and severity of acid-related symptoms after discontinuation of proton-pump inhibitor will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with typical reflux symptoms (heartburn and/or acid regurgitation) validated by standard questionnaire GerdQ.16
2. Aged from 18 to 70 years old.
3. Willing to receive H. pylori eradication therapy.

Exclusion Criteria:

1. Symptomatic reflux patients with high grade erosive esophagitis ( Los Angeles classification Grade C and D) or Barrett's esophagus documented by endoscopy.
2. Symptomatic reflux patients with a history of using PPI in recent one month.
3. Subjects with known allergy to PPI.
4. Peptic ulcer disease
5. Cancers of the esophagus, stomach, and duodenum
6. Esophageal or gastric varices
7. Active upper gastrointestinal bleeding within 7 days prior to enrollment
8. Status after total or subtotal gastrectomy
9. Pregnancy
10. Use of anticoagulants or antiplatelets within one week prior to enrollment
11. Subjects with bleeding tendency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive reflux patients documented by validated questionnaires (GerdQ) and upper endoscopy will be enrolled from the outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-09; Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of acid-related symptoms with GerdQ | 2 weeks after PPI
  To compare the incidence and severity of acid-related symptoms after discontinuation of proton-pump inhibitor between reflux patients with and without H. pylori infection

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chia Lee, MD,PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan